PRINCIPAL INVESTIGATOR: Scott Norberg, DO

**STUDY TITLE:** A Pilot Study of E7 TCR T Cell Induction Immunotherapy for Stage IIB-IVA

Cervical Cancer

STUDY SITE: NIH Clinical Center

Cohort: Treatment - Affected Patient

Consent Version: 11/4/2020

## WHO DO YOU CONTACT ABOUT THIS STUDY?

Principal Investigator: Scott Norberg, DO

Phone: 301-275-9668

Email: scott.nrorberg@nih.gov

#### KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you in making your decision about participating in this study. Additional information that may help you make a decision can be found in other sections of the document. Taking part in research at the NIH is your choice.

You are being asked to take part in this study because you have been diagnosed with Stage IIB-IVA cervical cancer. In addition, you completed the screening evaluation and were found to be eligible to take part in this research study.

The purpose of this study is to determine if E7 TCR cells can be given safely prior to your return to your cancer doctor for further treatment.

The use of E7 TCR T cells in this study is considered investigational, which means that it has not been approved by the U.S. Food and Drug Administration (FDA) to treat cervical cancer caused by HPV. However, the FDA has given us permission to use E7 TCR T cells in this study.

Standard treatment for your cancer consists of chemotherapy with radiation. Standard treatment is curative for most patients. However, some patients will have cancer recur at a new location after standard treatment, and when this happens it is not curable.

The goal of this study is to find out if it is possible to treat patients with your type of cancer with the experimental treatment (the E7 T cells) prior to getting standard treatment. We hope it will shrink the cancer and possibly prevent it from recurring at a new site later, but we do not know if this will be the case.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 11/4/2020


The experimental treatment is given before standard treatment and therefore will delay standard treatment. Your standard treatment may be delayed for up to 6 weeks after infusion of E7 TCR T Cells. It will require hospitalization, collection of a large volume of blood cells using a procedure called apheresis, biopsies of your tumor, and close follow up with visits to the NIH Clinical Center to monitor your cancer and the treatment side effects.

If your cells do not grow, you will not be able to receive the cell infusion. At the time we determine that your cells are not growing, we will inform you and discuss your options with you.

The single cycle of chemotherapy that is given as part of the experimental treatment has side effects that may include nausea, vomiting, diarrhea, hair loss, and decreased blood counts. These side effects are similar to the side effects you might experience from the standard chemotherapy you might receive even if you were not in this trial.

Also, as part of the experimental treatment, you will receive a drug called aldesleukin. The aldesleukin has side effects that may include fever, chills, low blood pressure, high heart rate, body swelling, and fatigue. Aldesleukin may have severe side effects that include lung failure, coma, and kidney failure. A complete list of side effects from the study medications is provided in this consent.

Being in this trial will not prevent you from receiving standard treatment for your cancer, although it will be delayed for up to 6 six weeks after the infusion of E7 TCR T Cells. If you do not want to delay standard treatment, or undergo any of the research procedures you may not want to join this trial. If you choose not to participate in this study you will receive standard treatment without the experimental treatment with your home oncologist.

You might wish to join this trial if you are willing to receive the experimental treatments and are interested in helping to find new ways to improve the treatment of this type of cancer.

If you decide to join this study, here are some of the most important things that you should know that will happen:

- You may only participate in this study if you have been diagnosed with Stage IIB-IVA cervical cancer. The primary treatment for this condition is chemoradiation. Unfortunately, not all patients are cured with this therapy.
- The therapy used in this study is called T cell therapy. Immune cells from your blood will be genetically modified in the laboratory to give them the ability to attack the human papillomavirus which causes cervical cancer.
- You completed the screening tests and you were found eligible for the study. If you decide to take part in this study, you will have a procedure to collect your T cells from the peripheral blood. These cells will be modified in the laboratory and will be given back to you by a one-time infusion into a vein. You will receive chemotherapy prior to getting the cells and a drug called aldesleukin afterwards. These drugs activate the gene-engineered T cells and help them proliferate. You will stay in the hospital for 2-3 weeks.
- You may experience side effects from taking part in this study. The most common side effects include decreased blood counts requiring transfusions, fevers, chills, nausea, low

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


blood pressure and high heart rate. It is possible that you could develop more serious, temporary, long-lasting or permanent side effects including death.

- We may draw your blood every day for research while you are in the hospital and we may ask you to have a cervical biopsy for research, about 6 weeks after the cell infusion.
- If you are a sexually active person capable of becoming pregnant, it is important that you do not become pregnant during your participation in this study. You must agree to use birth control from the time of enrollment on this study to four months after treatment.
- After the study follow-up period has ended, we would like to talk with you for 5 years to see how you are doing. We will ask you to participate in a long-term follow-up study where we will follow you for 15 years from the time you receive the cells.

Just as we do not know what side effects you might have, we cannot know if you may benefit from taking part in this study. If you do not benefit, this study and the results from our research may help others in the future.

You are free to stop participating in the trial at any time. If you decide to stop, the study doctor may ask you to agree to certain tests to make sure it is safe for you to stop.

The remaining document will now describe more about the research study. This information should be considered before you make your choice. Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

This is a research study. The purpose of this research study is to determine if E7 TCR T cells can be given without delaying your standard treatment whether that is surgery or radiation therapy with chemotherapy unless that delay is because the therapy is shrinking your tumor(s). We hope this treatment will shrink the cancer and possibly prevent it from recurring at a new site later, but we do not know if this will be the case.

We are asking you to join this research study because you have been diagnosed with Stage IIB-IVA cervical cancer. In addition, you completed the screening evaluation and were found to be eligible to participate in this research study.

We have developed an experimental therapy that involves taking white blood cells called lymphocytes from you, growing them in the laboratory in large numbers, genetically modifying them to give them new genes (T Cell Receptor (TCR)), which help them recognize the cancer, and

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


then giving the cells back to you. In this study, we are modifying your white blood cells with a retrovirus that has the gene for a TCR that recognizes the HPV-16 E7 protein. So far, the HPV-16 E7 has been found only on tumor cells. This type of treatment is called cell therapy. We have given these cells to patients in a previous clinical trial where the goal was to find the most effective yet safe dose of E7 TCR T cells.

Before receiving the E7 TCR cells, you will receive 2 FDA approved chemotherapy drugs to temporarily suppress the immune system to improve the chances that the experimental cells will be able to survive in the body. After the cells are given, you will receive aldesleukin (IL-2) to help these cells stay alive longer. Once you have completed this therapy, you will be seen in our clinic to see if your cancer has grown and whether you are recovering from any toxicities experienced during the trial. If your cancer is getting smaller we will continue to see you in clinic. If your cancer doesn't get smaller or goes away completely you will be referred back to your home oncologist for standard treatment.

#### WHAT WILL HAPPEN DURING THE STUDY?

## Before you begin study therapy

You will need to supply an updated complete list of your current medications to the study doctor. This includes over-the-counter medications and herbal supplements. Some medications may interfere with the study drugs and it is important that your study doctor and prescribing physician be aware of any potential risks so that they can prescribe alternative medications as necessary. If you do not already do so, please carry a list of your medications at all times.

This study has several stages after screening:

| Stage | Timeframe | Location | Comments & Instructions |
|---|---|---|---|
| Baseline | Within 30 days prior to leukapheresis | Inpatient or outpatient | Complete physical examination, vein assessment, blood tests |
| Baseline | Within 4 weeks<br>prior to starting<br>chemotherapy<br>regimen | Inpatient or outpatient | Clinical staging (may include CT scan, MRI scan, PET scan), tumor measurements, optional tumor biopsy (any time prior to chemotherapy), Chest x-ray, ECG, Cardiac and/or pulmonary testing |
| Leukapheresis<br>before<br>treatment | At least 11 days<br>prior to cell<br>infusion | Inpatient or outpatient | This is a half to full day appointment. |
| Chemotherapy (day -6 to -2) | 1 week | Inpatient | Receive IV chemotherapy to prepare your immune system for the cells. |

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


| Stage | Timeframe | Location | Comments & Instructions |
|---|---|---|---|
| Cells and aldesleukin (Day 0-2) | 1-3 days | Inpatient and possibly ICU | Receive 30 billion E7 TCR cells IV and then high dose aldesleukin about every 8 hours for up to 6 doses. |
| Recovery | 1-2 weeks | Inpatient unit | Recover from the effects of treatment. |
| Follow -up | 3 weeks and 6 weeks post cell infusion. All patients will be referred for standard of care treatment 6 weeks after E7 TCR cell infusion. | Outpatient | 3 weeks post E7 TCR cell infusion: Return to clinic for physical exam, labs, review of side effects. 6 weeks post E7 TCR cell infusion: Return to clinic for physical exam, review of side effects, labs, scans, optional tumor biopsy. |

#### **Baseline**

Prior to receiving the experimental treatment, you will have additional tests. These may include imaging procedures, and laboratory tests. You will also have a large catheter inserted into a vein so that leukapheresis can be performed (see below). You may be admitted to the hospital for these tests and procedures.

## **During study therapy**

## Cell harvest and growth

You will have a procedure called leukapheresis to obtain white blood cells from you. These cells will be grown in the lab and genetically modified to recognize a protein on your tumor cells. You may have enrolled on protocol 16C0061 to undergo leukapheresis. If you had a leukapheresis procedure and we have collected cells, then you will not need to do it again.

If your cells do not grow, you will not be able to receive the cell infusion. If that happens, we will look at alternative experimental treatments at the NIH Clinical Center or refer you to the care of your referring home physician. We usually know after about 2 weeks whether the cells will grow well enough to be used as an experimental treatment on this protocol. At the time we determine that your cells are not growing, we will inform you and discuss your options with you.

## Leukapheresis

Leukapheresis is a procedure that allows us to remove certain types of blood cells from you and return the rest of your blood. It is a very common procedure that is done routinely here at the NIH with very few risks. During leukapheresis, blood is removed from you through a needle in your arm, circulated through a machine that divides whole blood into red cells, plasma (the liquid component of blood), and leukocytes (or white cells), and then the plasma and red cells are returned

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


to you through a second needle in your other arm. If the procedure cannot be done through a needle in your arm, a central catheter may need to be placed. The white blood cells may be used to help grow your anticancer cells. In addition to the leukapheresis, we will also ask you to undergo one additional apheresis procedure around 4 weeks after your cell treatment to see how this therapy affects your immune system and see if cells we gave you are still active.

#### **Intravenous Catheter**

To receive this treatment, you may need to have a central venous catheter. This catheter is placed under the skin and enters a major vein. The area will be numbed with an anesthetic before the catheter is put in. The procedure will be discussed with you in detail prior to the catheter placement.

#### **Blood Draws**

Blood will be drawn frequently during your treatment. Most of the blood draws will be to monitor your health during and after the lymphocyte infusion. During that time, we will remove between 1 and 9 teaspoons of blood daily to study the effects of the treatment regimen on your immune system. If you experience side effects in your kidneys, we will collect 1 additional teaspoon of blood. In addition, some blood samples will be drawn for research purposes. The maximum amount of blood for research is approximately 2.3 cups in 8 weeks. Additional blood draws might be necessary to investigate T cell responses and serum cytokine levels in cases of clinical events such as rapid progression of malignancy or side effects. These samples will be used to study how your immune system is affected by the cell therapy. Some of the samples may be used for other or future research conducted by the investigational team or other researchers.

## Chemotherapy Regimen (Day -6 through Day -2)

After we have grown the E7 TCR cells to large numbers in the laboratory, you will be admitted to the hospital to begin your experimental treatment. You will be given two chemotherapy medicines, cyclophosphamide and fludarabine, to make space in your immune system so the E7 TCR cells can work without any interference from the cells in your immune system. These medicines may cause your tumor to shrink some, but this shrinkage is anticipated to be only partial and of small duration. The main purpose of the chemotherapy is to see if we can make the cells more effective in fighting cancer tumors. Animal experiments have indicated that chemotherapy can make the infused cells more effective in fighting your cancer, but it is not known whether this is true in humans. The cyclophosphamide will be given into your catheter over 1 hour for two days (Day -6 and Day -2) and the fludarabine will be given into your catheter for 30 minutes every day for five days (Day -6 through Day -2). The side effects of these medicines are described on the following pages. To decrease your risks for getting certain infections, we will treat you with medications that work against bacteria, virus, and, if needed, ones that work against fungal infections. You will have to take these for 6 months or longer, depending on the recovery of your infection fighting blood cells.

#### Cell Infusion and Aldesleukin Regimen (Day 0 through Day 2)

You will be given 30 billion cells through the IV over 20-30 minutes one to four days after the last dose of chemotherapy. Within 24 hours after your cell infusion you will be given high dose aldesleukin through one of the IVs. It will be given as a 15-minute infusion about every 8 hours

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


 IRB APPROVAL DATE: 01/02/2021

IRB NUMBER: 20C0116

for up to five days after the cell infusion. Aldesleukin is a cell growth factor and it is thought that it will help the cells live longer in your body.

The day after your cells are infused, we may give you G-CSF (filgrastim) as a shot or injection under the skin every day to stimulate your blood cells until they increase to a sufficient number to help you fight infections. We will watch you closely during this entire time for any side effects of this experimental regimen. We will discuss the side effects below and we will include in your care all the medicines and treatments to prevent as many of these side effects as we can and to make you as comfortable as we can.

## When you are finished with the T cell treatment

## Recovery

You will recover in the hospital until you are well enough to go home. This will likely take 7-12 days after you have received cells; however, you may need to stay in the hospital longer until you are well enough to go home. We will continue to give you supportive medications, do laboratory tests, and watch you closely for any side effects until we feel your condition is stable.

In addition to the laboratory tests to monitor your condition, we will remove between 1 and 9 teaspoons of blood daily to study the effects of this regimen on your immune system. If you experience side effects in your kidneys, we will collect 1 additional teaspoon of blood and about 6 teaspoons of urine to help us determine the cause of these side effects. The maximum amount of blood for research is approximately 2.3 cups in 8 weeks.

# Follow up and Evaluation of Experimental Regimen

You will need to come for a clinic visit approximately 3 weeks (21 days) after cell administration for a physical examination and blood work. If your tumor appears to be growing, we will refer you back to the care of your home physician. If not, you will need to come for a clinic visit again at 6 weeks (42 days) after your cell administration to see how your tumor is responding to the treatment. Regardless of the response to treatment, you will then be referred back to your home physician for further care after the 6 week visit.

At the 3 week visit, you will have lab tests and a physical examination performed. This visit is to make sure you are recovering from the treatment. At the 6 week response assessment visit, you will have lab tests, imaging studies and a physical examination. At one of your follow up visits, you may undergo apheresis or have about 8 tubes of blood drawn (4 tablespoons) so that we can see the effect this therapy had on your immune system and if the cells we gave you are still alive.

## Gene Therapy Long Term Follow up

You will be followed on a separate protocol once you finish the cell therapy. We will ask you to sign a separate consent for this other protocol. Because we do not know the long-term side effects of gene therapy, we will ask you to take part in long term follow up for the next 15 years. The Food and Drug Administration (FDA) requires that people who receive gene therapy be watched even after they complete the study. We will ask you questions about your health and ask you to have a physical exam every year. We will also collect your blood over the next several years. If you return to your home physician after treatment here, we will ask you to have them send us a copy of your physical exam and your blood samples. We will collect blood samples right after you receive the cells, and at 3, 6 and 12 months after treatment, and then every year after that (2

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


teaspoons each time) up to 5 years. This testing will help us learn if the cells have grown or changed in your body. For this reason, we ask that you continue to provide us with a current address and telephone number, even after you complete this research study.

At the time of your death, no matter the cause, we may request consent from your family for an autopsy. This will allow us to obtain important information about the safety of this experimental treatment. Please discuss this with your family to inform them of this potential request.

#### HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this study, your involvement will last for up to 5 years:

• After you receive E7 T cells, you will be seen in the clinic at 3 weeks and 6 weeks post cell infusion. After the 6 week visit, you will be referred back to your home doctor to receive standard of care definitive treatment. We will then contact you once a year to ask you questions about your disease and any treatments for the disease that you have received. This will happen for a total of 5 years.

Your involvement on the Gene Therapy Long Term Follow Up Study will be 15 years once you receive the E7 T cells.

#### HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

Not everyone screened for the study will be eligible to receive study therapy. It is expected that up to 18 people may receive study therapy in this study.

## WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

The risks and discomforts of this research study can be significant. This experimental treatment can lead to long-term decrease in your immune function. It is also possible that you may lose your fertility following this experimental treatment. It is possible, although unlikely, that this experimental treatment may cause your death.

We will discuss the side effects of this experimental treatment with you. You will be given medicines, transfusions, and treatments to prevent or treat the side effects including drugs to prevent and/or treat different types of infections. We will try to make you as comfortable as possible.

## **Blood samples**

Side effects of repeated blood sampling depend in part on how the blood is drawn. If through a central venous catheter, risks include contamination of the catheter which would result in a serious blood stream infection, requiring admission to the hospital and giving you antibiotics through the vein; if blood is drawn through a needle into your skin, side-effects could include pain and bruising in the area where the blood was drawn. Other side-effects can include bruising, redness, discomfort or bleeding at the site of the needle stick, and possible lightheadedness, or rarely, fainting. If you have too much blood taken over a prolonged period, your red blood cell count may drop (this is called "anemia"). As a precaution, we will check your red blood cell level, and give you iron treatment or a blood transfusion if needed.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


## Leukapheresis

During the leukapheresis procedure, you may have some tingling in your face and lips due to the medicine used to keep your blood from clotting during the procedure. The nurses may give you a calcium-containing antacid to chew that takes away this tingling. Rarely, people may experience lightheadedness or dizziness. We ask that you eat prior to the procedure to prevent this. Rare complications of this procedure are lowered blood pressure, bleeding or bruising where the needles are put in your arms.

#### Administration of E7 T cells

The cells we will be giving you have a type of virus (retrovirus) put into them that recognizes the HPV E7 protein. Although this retrovirus is not active, there is the rare possibility that it may cause infection. The cells could also cause you to develop another type of cancer, such as leukemia or lymphoma. These specific gene-modified cells have been given before but we do not have much information about the side effects.

#### Potential risks include:

- Fever, chills and shortness of breath, which may last for a few hours (common)
- Lung congestion causing shortness of breath
- Severe reaction to the cells which would include very low blood pressure and damage to your heart, lung, and/or kidneys
- As this is a new experimental therapy which has been given to only a few patients, side effects that we do not anticipate that may cause your condition to deteriorate may be encountered. Any new information that becomes available during the course of this study will be shared with you.
- A patient treated with E7 TCR T cells on another protocol, who had breathing problems from advanced cancer in the lungs, developed severe breathing, blood pressure, and kidney toxicity that required temporary support with a breathing machine, blood pressure medicines, and dialysis and this resulted in injury to her toes and feet.
- Another patient treated with E7 TCR T cells on another protocol developed confusion and low blood pressure after E7 TCR T cells and one dose of aldesleukin that required a breathing machine, blood pressure medicine and dialysis. The patient also developed an inflammatory disorder characterized by fevers, prolonged low blood counts, and abnormal blood tests for inflammation that resolved following treatment with steroids. The patient also had delayed recovery of blood counts that was caused by prior chemotherapy, prior pelvic radiation and poor nutrition.
- You will be treated on this gene transfer protocol with a viral vector that was manufactured at the NCI Surgery Branch Vector Production Facility before May 2016. An internal review of the facility that made the vector for this protocol determined that the facility needed to be closed due to manufacturing issues. We know of no additional risks related to the previously produced vector for patients who have received cells with vectors made in this facility as the vectors were extensively tested by outside experts. Therefore, the IRB has determined that the potential benefit to you outweighs the potential risks.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# Other study drugs

The side effects of cyclophosphamide, fludarabine, high dose aldesleukin and some of the other medications you will receive are listed below:

## Potential side effects from aldesleukin

| Likely | Less Likely | Rare but Serious |
|---|---|---|
| <ul> <li>Fever, chills, and fatigue</li> <li>Lowered platelet and red blood cell levels that may require transfusions</li> <li>Significant fluid retention causing weight gain (as much as 20 pounds).</li> <li>Low blood pressure</li> <li>Increased heart rate</li> <li>Low urine output</li> <li>Swelling in your extremities</li> <li>Fluid in your lungs that can require oxygen</li> <li>Dry mouth, nausea, vomiting and diarrhea;</li> <li>Rash, itching; and changes in skin or hair pigmentation, called vitiligo;</li> <li>Changes in mental status, including confusion, difficulty sleeping or vivid dreams; this can be severe and require sedation and monitoring in the ICU</li> </ul> | <ul> <li>Decrease in thyroid function that may require daily thyroid hormone replacement;</li> <li>Abnormal kidney and liver function that can be severe;</li> <li>Abnormal heartbeats or low blood pressure that may require treatment in the ICU.</li> <li>Breathing problems which may need monitoring in ICU and insertion of a breathing tube.</li> </ul> | <ul> <li>Bowel perforation (a hole) requiring longer hospitalization or surgery.</li> <li>Autoimmune disease, where your immune system attacks cells in organs of your body. Should this occur, you will be treated with steroids to stop the immune response.</li> <li>Damage to the heart muscle or heart attack</li> <li>Loss of blood flow to the extremities due to medicines used to treat very low blood pressure and shock. In one instance a patient had to have her lower arm amputated after treatment with these medicines.</li> <li>Aldesleukin is mixed with human albumin which could cause an allergic reaction or potentially transmit viral infections, although we have not had this occur.</li> </ul> |

# Potential side effects from cyclophosphamide and fludarabine

| Likely | Less Likely | Rare but Serious |
|---|---|---|
| <ul> <li>Changes in blood counts<br/>including: low red cell<br/>count (causing fatigue<br/>and shortness of breath),<br/>low platelet count<br/>(increasing the risk of</li> </ul> | <ul><li>Bleeding</li><li>Infection</li><li>Bladder irritation with<br/>bloody urine</li></ul> | <ul> <li>Heart damage</li> <li>Lung damage</li> <li>Kidney damage</li> <li>Inflammation of the eye resulting in blindness</li> </ul> |

# PATIENT IDENTIFICATION

# Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


bleeding and bruising), decrease in white blood cells (increasing the risk of infection and the need for treatment with antibiotics or other treatment)

- Loss of appetite, nausea, vomiting,
- Diarrhea, stomach pain
- Mouth sores
- Hair loss
- Fatigue
- Muscle or joint aches

- Severe allergic reaction (difficulty breathing/swelling)
- Headache or dizziness
- Sweating
- Swelling of arms or legs
- Skin changes, rash, blisters
- Weakness
- Hearing loss

- Inflammation of nervous system resulting in death
- Epstein Barr Virus
  Lymphoma. This can be
  fatal (Two patients on
  other studies in the
  Surgery Branch
  developed EBV
  lymphoma, and one died
  as a result of this
  disease.)
- Loss of fertility
- Death due to complications resulting from suppression of the immune function.

## Gene Therapy Risk of Cancer and Other Diseases

We are unsure if this type of gene therapy will cause you to become sick in the future. It is possible that it may cause your immune system or nerves not to work well or cause a sickness of your blood cells or even a cancer (for example leukemia). We do not know if you will develop any of these disorders, but you need to be aware of this possible risk. Children in France and England received gene therapy for a particular disease of the immune system. Most of the children were cured but 5 children out of 22 later developed leukemia and one died. Experts who looked at these cases thought that the gene therapy caused the leukemia in these children. To watch you for this risk we will be testing your blood as described before.

# **Biopsies**

Biopsy of the primary tumor is optional and may be performed before getting the cells and approximately 6 weeks after T cell injection(s). They will be done using local anesthesia by a gynecologist doctor. In some cases where the tumor cannot be seen using the instruments in the clinic, you might have the biopsy performed in the operating room under general anesthesia. Risks associated with the biopsies are pain and bleeding at the biopsy site. Although rare, serious risks associated with general anesthesia include an adverse drug reaction, stroke, heart attack or death. You will be asked to sign a separate consent prior to each procedure involving anesthesia.

#### X-ray examination

An x-ray examination exposes you to a small amount of radiation, corresponding to one-fifth of the dose a person gets each year from natural sources, such as the sun and the ground. This small amount of radiation is not considered dangerous.

#### CT scan, MRI and PET

During a CT scan, and PET, you're briefly exposed to much more radiation than you would be during a plain X-ray. Radiation exposure potentially increases your risk of developing cancer. Although rare, the intravenous (IV) contrast material involved in some CT, PET and MRI scans causes medical problems or allergic reactions in some people. Most reactions are mild and result

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


in hives or itchiness. In rare instances, an allergic reaction can be serious and potentially life threatening. Make sure to tell your study doctor if you've ever had a prior reaction to contrast material during medical tests.

Risks for gadolinium enhanced MRI scans:

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis" which has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is not normal or if you received gadolinium within the previous month.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA recently issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. Some types of gadolinium contrast drugs are less likely to remain than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain.

#### What are the risks of radiation from being in the study?

During your participation in this research study, you will be exposed to radiation from a CT scan, PET, or CT-guided biopsy. The amount of radiation exposure you may receive from these procedures is equal to approximately 6.2 rem. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." This study will expose you to more radiation than you get from everyday background radiation. No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The PET and CT that you get in this study will expose you to the roughly the same amount of radiation as 20.7 years' worth of background radiation. Being exposed to too much radiation can cause harmful side effects such as an increase in the risk of cancer. The risk depends on how much radiation you are exposed to. Please be aware that about 40 out of 100 people (40%) will get cancer during their lifetime, and 20 out of 100 (20%) will die from cancer. The risk of getting cancer from the radiation exposure in this study is 0.6 out of 100 (0.6%) and of getting a fatal cancer is 0.3 out of 100 (0.3%).

#### **Radiation Exposure in People Capable of Becoming Pregnant**

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


Page **12** of **20** 

You may not participate in this study if you are pregnant. If you are able to become pregnant, we will perform a pregnancy test before exposing you to radiation. You must tell us if you may have become pregnant within the previous 14 days because the pregnancy test is unreliable during that time.

#### **Intravenous Catheter**

The risks associated with placing some catheters include pain, bleeding, infection and collapsed lung. Lung collapse is treated by putting a tube into your chest for a few days to allow your lung to expand. Pressure is placed on any area that might bleed. Other IVs may be needed in one or both of your arms if we need to give you extra fluids, medicines, or nutrition. The long-term risks of the catheter include infection and clotting of your veins. If these occur, it may be necessary to remove the catheter. These risks will be explained to you in more detail at the time of insertion.

# What are the risks related to pregnancy?

If you are able to become pregnant, we will ask you to have a pregnancy test before starting this study. You will need to practice an effective form of birth control before starting study treatment, during study treatment, and for 4 months after you finish study treatment (the restricted period).

Effective forms of birth control may include:

- Abstinence
- Intrauterine device (IUD)
- Hormonal (birth control pills, injections, or implants)
- Tubal ligation
- Vasectomy

If you become pregnant, there may be unknown risks to the fetus or unborn child, or risks that we did not anticipate. There may be long-term effects of the treatment being studied that could increase the risk of harm to a fetus. You must tell the study doctor if your birth control method fails during the restricted period. If you think or know you have become pregnant during the restricted period, please contact the study team as soon as possible.

# WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You might not benefit from being in this study.

However, the potential benefit to you might include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer.

## Are there any potential benefits to others that might result from the study?

In the future, other people might benefit from this study because the knowledge gained from this study may help in developing treatments for those who have cervical cancer.

## WHAT OTHER OPTIONS ARE THERE FOR YOU?

Before you decide whether or not to be in this study, we will discuss other options that are available to you. Instead of being in this study, you could:

choose to be treated with surgery, radiation or with drugs already approved by the FDA for your disease

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


- choose to take part in a different study, if one is available
- choose not to be treated for cancer but you may want to receive comfort care to relieve symptoms.

You should discuss with your doctor your other choices and their risks and benefits.

#### **DISCUSSION OF FINDINGS**

## New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

#### Return of research results

We do not plan to return research results to you. A summary of the research results will be posted on Clinicaltrials.gov at completion of the study.

## EARLY WITHDRAWAL FROM THE STUDY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease worsens or comes back during treatment
- if you have side effects from the treatment that your doctor thinks are too severe
- if you become pregnant
- if new information shows that another treatment would be better for you
- if you do not follow the study rules
- if the study is stopped for any reason

In this case, you will be informed of the reason therapy is being stopped.

After therapy is stopped we would like to see you for a safety visit approximately 21 days after your last dose.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to our collaborators or designated representatives.

# STORAGE, SHARING AND FUTURE RESEARCH USING YOUR SPECIMENS AND DATA

#### Will Your Specimens or Data Be Saved for Use in Other Research Studies?

As part of this study, we are obtaining specimens and data from you. We will remove all the identifiers, such as your name, date of birth, address, or medical record number and label your specimens and data with a code so that you cannot easily be identified. However, the code will

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


Page **14** of **20** 

be linked through a key to information that can identify you. We plan to store and use these specimens and data for studies other than the ones described in this consent form that are going on right now, as well as studies that may be conducted in the future. These studies may also be done on protocol 16C0061 if you are co-enrolled on that study. These studies may provide additional information that will be helpful in understanding cervical cancer, or other diseases or conditions. This could include studies to develop other research tests, treatments, drugs, or devices, that may lead to development of a commercial product by the NIH and/or its research or commercial partners. There are no plans to provide financial compensation to you if this happens. Also, it is unlikely that we will learn anything from these studies that may directly benefit you.

I give permission for my coded specimens and data to be stored and used for future research as described above.

| Yes | No |
|----------|----------|
| Initials | Initials |

## Will Your Specimens or Data Be Shared for Use in Other Research Studies?

We may share your coded specimens and data with other researchers. If we do, while we will maintain the code key, we will not share it, so the other researchers will not be able to identify you. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at NIH, other research centers and institutions, or commercial entities.

I give permission for my coded specimens and data to be shared with other researchers and used by these researchers for future research as described above.

| Yes | No |
|----------|-----------------|
| Initials | <b>Initials</b> |

If you change your mind and do not want us to store and use your specimens and data for future research, you should contact the research team member identified at the top of this document. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy your specimens and data. For example, if some research with your specimens and data has already been completed, the information from that research may still be used. Also, for example, if the specimens and data have been shared already with other researchers, it might not be possible to withdraw them.

In addition to the planned use and sharing described above, we might remove all identifiers and codes from your specimens and data and use or share them with other researchers for future research at the NIH or other places. When we or the other researchers access your anonymized data, there will be no way to link the specimens or data back to you. We will not contact you to ask your permission or otherwise inform you before we do this. We might do this even if you

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


answered "no" to the above questions. If we do this, we would not be able to remove your specimens or data to prevent their use in future research studies, even if you asked, because we will not be able to tell which are your specimens or data.

NIH policies require that your clinical and other study data be placed in an internal NIH database that is accessible to other NIH researchers for future research. These researchers will not have access to any of your identifiers, such as your name, date of birth, address, or medical record number; and your data will be labeled with only a code. We cannot offer you a choice of whether your data to be placed in this database or not. If you do not wish to have your data placed in this database, you should not enroll in this study.

# How Long Will Your Specimens and Data be Stored by the NIH?

Your specimens and data may be stored by the NIH indefinitely.

# Risks of Storage and Sharing of Specimens and Data

When we store your specimens and data, we take precautions to protect your information from others that should not have access to it. When we share your specimens and data, we will do everything we can to protect your identity, for example, when appropriate, we remove information that can identify you. Even with the safeguards we put in place, we cannot guarantee that your identity will never become known or someone may gain unauthorized access to your information. New methods may be created in the future that could make it possible to re-identify your specimens and data.

## COMPENSATION, REIMBURSEMENT, AND PAYMENT

# Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

# Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

On this study, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy. You will be given a summary of the policy which provides more information.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

 If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

## **CONFLICT OF INTEREST (COI)**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

The National Institutes of Health and the research team for this study are using E7 TCR (biological product) developed by Center for Cancer Research through a joint study with your study team and Kite Pharma. This means it is possible that the results of this study could lead to payments to NIH. By law, the government is required to share such payments with the employee inventors. You will not receive any money from the development of E7 TCR.

Kite Pharma will provide financial support for this study.

#### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

#### Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor (Center for Cancer Research) or their agent(s)

When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you

#### PATIENT IDENTIFICATION

## Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

If we share your specimens or data with other researchers, in most circumstances we will remove your identifiers before sharing your specimens or data. You should be aware that there is a slight possibility that someone could figure out the information is about you.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

## **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

# **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical information that we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


#### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

# PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Scott Norberg, DO, <a href="mailto:scott.norberg@nih.gov">scott.norberg@nih.gov</a>, 301-275-9668. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

#### **CONSENT DOCUMENT**

Please keep a copy of this document in case you want to read it again.

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


| Adult Research Participant: I have read the exto discuss it and to ask questions. I consent to pa | | given the opportunity |
|---|---|---|
| Signature of Research Participant | Print Name of Research Participant | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| Witness to the oral short-form consent proces | ss only: | |
| Witness: | | |
| Signature of Witness* | Print Name of Witness | Date |
| *NIH ADMINISTRATIVE SECTION TO INTERPRETER: An interpreter, or other individual, who speed the administration of informed consent and servals also serve as the witness. An interpreter, or other individual, who speed the administration of informed consent but did reproviding interpretive support is: | aks English and the participant's preferred ved as a witness. The investigator obtain aks English and the participant's preferred | I language facilitated ing consent may not I language facilitated |

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1) Version Date: 11/4/2020


